CLINICAL TRIAL: NCT05145738
Title: Pilot Testing a Computer Delivered Tobacco Cessation Intervention in Outpatient Clinical Settings: A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00300496
Record Dates: First submitted 2021-11-23; First posted 2021-12-06 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Tobacco Smoking
MeSH Terms: conditions — Tobacco Smoking

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Care providers, investigators and outcome assessors will be blind to avatar versus no avatar conditions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- C-Raven + Avatar (Experimental): Computer delivered intervention with Avatar as virtual counselor plus linkage to community health worker
  Interventions: Behavioral: C-Raven with avatar
- C-Raven (Active Comparator): Computer-delivered intervention without virtual counselor, with linkage to community health worker
  Interventions: Behavioral: C-Raven without avatar

INTERVENTIONS:
Behavioral: C-Raven with avatar — Computer delivered intervention with the investigators' avatar; with linkage to community health worker.
  Arms: C-Raven + Avatar
Behavioral: C-Raven without avatar — Computer delivered intervention without the investigators' avatar; with linkage to community health worker.
  Arms: C-Raven

SUMMARY:
The investigators have developed a hybrid computer- and person-delivered intervention, called "C-Raven" for smoking cessation that is tailored to people with tobacco use in Baltimore City. The computer delivered component consists of two ~20 minute sessions on an iPad guided by Edna Poe, an interactive avatar. These sessions are followed by elective in vivo initiation of nicotine replacement therapy (NRT). Community health workers (CHWs) trained in smoking cessation and motivational interviewing provide 6 weeks of supportive follow up counseling. The investigators propose a pilot of the intervention package in the Tobacco Treatment and Lung Cancer Screening Clinic (TTLCSC) at Johns Hopkins Hospital, and the Johns Hopkins Broadway Center for Addiction, assessing feasibility and acceptability of using this tool in these clinical settings. In addition, the investigators will compare whether the use of a virtual counselor is associated with greater satisfaction and engagement with the program.

To this end, the investigators propose a two-arm randomized controlled trial, randomizing up to 90 individuals with tobacco use to the current CRAVEN program which includes a virtual counselor, to CRAVEN without a virtual counselor. Primary outcomes include intervention feasibility and acceptability. The investigators will secondarily examine uptake and maintenance of pharmacotherapy for tobacco cessation, readiness to quit smoking, and tobacco cessation (7 day abstinence) at 6 months, patient satisfaction by intervention arm and CHW engagement by intervention arm.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age receiving care in one of the two specified clinics
* Current daily smoker and has smoked >100 cigarettes in their lifetime
* English speaking
* Cognitively able to understand proposed research design

Exclusion Criteria:

* Actively psychotic or other severe mental health symptoms
* Any contraindication to NRT use
* Hearing impaired (unable to listen to audio component of intervention)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-12-23 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Percent of persons agreeing to participate among those referred | 3 months
  Feasibility will be assessed with percent of persons agreeing to participate among those referred.
Percent of contacts made with community health worker | 3 months
  Implementation will be assessed with percent of contacts made with community health worker.

SECONDARY OUTCOMES:
Readiness to quit smoking as assessed by a visual analog scale | Immediately post intervention
  A visual analog scale of 0-100 with 0 indicating not ready to change and 100 indicating ready to change.
Uptake of pharmacotherapy as assessed by a yes/no response | 3 months
  Any uptake of nicotine replacement therapy or varenicline or wellbutrin. Dichotomous yes/no response will be collected.
Smoking cessation as assessed by 7-day no tobacco use self report | 3 months
  7 day point prevalence abstinence. No tobacco use for 7 days by self report - yes/no.

CONTACTS AND LOCATIONS:
Overall Officials: Geetanjali Chander, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Tobacco Treatment Clinic at Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No